CLINICAL TRIAL: NCT01936753
Title: The Impact of Mentor Mother Programmes on PMTCT Service Uptake and Retention at Primary Healthcare Facilities in Nigeria
Brief Title: The Impact of Mentor Mothers on PMTCT Service Outcomes in Nigeria
Acronym: MoMent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Human Virology, Nigeria (Other)
Collaborators: University of Maryland (Other); Federal Ministry of Health, Nigeria (Other Government)
Responsible Party: Principal Investigator, Dr. Nadia Sam-Agudu, Senior Techical Advisor, Pediatric and Adolescent HIV, Institute of Human Virology, Nigeria
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IHVN_WHO_PMTCT_MoMent; RPC531 (Other Grant/Funding Number: World Health Organization)
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: HIV
Keywords: PMTCT; HIV; Mentor Mothers; Nigeria; Retention; Adherence

STUDY DESIGN:
Intervention Model Description: This is a prospective paired cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mentor Mother Peer Support (Experimental): This is an enhanced behavioral intervention. Mentor Mothers trained with a standard study curriculum are assigned to pregnant HIV-positive women accessing care at Primary Healthcare Centers in study communities. Under close daily supervision, Mentor Mothers provide support and counseling for the mother-infant pairs until the exposed infant is 12 months old. Study participants in this arm also receive standard of care PMTCT services.
  Interventions: Behavioral: Trained Mentor Mother and Supervisor
- Routine Peer Support (No Intervention): Pregnant HIV-positive women receive standard-of-care PMTCT services (drugs, appointments, tests). These women are, per routine, assigned peer counselors who are also HIV-positive women with PMTCT experience but who do receive little or no standardized formal training, and are not closely supervised.

INTERVENTIONS:
Behavioral: Trained Mentor Mother and Supervisor — Trained, closely supervised Mentor Mothers guide and support the mother-infant pair to achieve timely and complete access to, and retention in PMTCT services along the entire cascade.
  Arms: Mentor Mother Peer Support

SUMMARY:
Nigeria has significant challenges in the delivery and coverage of PMTCT (Prevention of mother-to-child transmission of HIV) services. Only 30% of pregnant women living with HIV are provided anti-retroviral drugs for PMTCT. Less than 10% of HIV-exposed infants receive HIV testing for early diagnosis by age 2 months. Furthermore, an unacceptably high number of women with HIV who are enrolled in PMTCT programs do not complete them. In other words, uptake and retention in PMTCT programs in Nigeria is not adequate. Ultimately, mother-to-child transmission of HIV is high, resulting in a high number of new child HIV infections.

Mentor Mothers (MMs) are women living with HIV who provide peer support to other HIV-positive women. MM programs have been incorporated into PMTCT programs in several African countries with some success, but with varying levels of MM training and program structure. The MoMent (MOther MENTor) study investigates whether highly-structured MM programs will further improve uptake and successful completion of PMTCT services (eg testing and appointments) in Nigeria. The study also evaluates the impact of structured MM programs on other outcomes, including facility deliveries, new infant HIV infections, infant survival and maternal viral suppression. Rural areas are the focus of this study because of their particularly poor performance in PMTCT coverage and outcomes.

DETAILED DESCRIPTION:
Nigeria has had a national HIV/AIDS care and treatment program in place since 2003. Included in this national program are prevention programs; the largest of which is the prevention-of-mother-to-child transmission (PMTCT) program. Despite more than 10 yrs of providing PMTCT, Nigeria still has significant problems with uptake of, and retention in these services. Only 30% of HIV-positive pregnant women receive HIV drugs for both treatment and prophylaxis, and Nigeria has an estimated 41,000 new child infections annually, the highest of any country in the world.

Mentor Mothers (MM) are women living with HIV who are experienced users and navigators of HIV services, particularly PMTCT. Public health interventions engaging MM to support other HIV-positive women for linkage and retention in PMTCT and treatment services has been tested in South Africa, and has been adopted and applied in several other African countries. Similar MM programs have also been adopted and implemented in Nigeria since 2007; however, objective evaluations of MM impact on PMTCT service uptake and retention have not been performed to date.

While MM and similar peer support interventions have shown some success in other African countries, their implementation between and within countries has not been standardized. Incremental impact may be gained with more structured, objective-specific MM programming and service delivery.

The MoMent (MOther MENTor) is an implementation research study that is evaluating the impact of structured vs routine peer support on PMTCT outcomes in Nigeria, focusing on two North-Central states, the Federal Capital Territory and Nasarawa. The intervention consists of a simple but detailed standardized training curriculum for MMs coupled with daily MM supervision by dedicated personnel as well as standardized, user-friendly tools for both MMs and their supervisors to use for service delivery. These trained MM, along with trained MM Supervisors, form the basis of the Mentor Mother Intervention package. The choice of rural areas served by Primary Healthcare Centers is due to the fact that PMTCT coverage and uptake is lowest in these areas; the study sites are located in hard-to-reach-areas where a significant number of PMTCT-eligible clientele live.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and HIV-positive
* 15 years of age and above

Exclusion Criteria:

* Working or ever worked as a Mentor Mother
* Presenting in labor
* Does not plan to continue receiving services at study site

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only HIV-positive pregnant females are eligible for recruitment. All infants born live to these females are also enrolled.
Enrollment: 497 (Actual)
Dates: Start 2014-04-24 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Proportion of HIV-exposed infants presenting for DNA PCR testing by 2 months of age. | At 2 months (62 days) of age for the HIV-exposed infant.
  Early infant diagnosis (EID) is defined as the collection and processing of an HIV DNA PCR test for an HIV-exposed infant by 2 months of age. EID is done to ensure that HIV-positive infants will be promptly enrolled into HIV treatment programs and can start lifesaving Antiretroviral Therapy (ART) in timely fashion.
Proportion of HIV-positive mothers retained in PMTCT care at 6 months post-delivery. | At 180 days (6 months) post-delivery
  Maternal retention is determined by evaluating for at least 1 clinic visit made for each 30-day period for the first 180 days postpartum. The proportion of women making at least 3 of 6 monthly appointments are designated retained; this proportion is calculated for each study arm.

SECONDARY OUTCOMES:
Maternal viral suppression at 6 months postpartum | 6 months (169 to 197 days) post-delivery
  Proportion of HIV-positive mothers with undetectable viral load (<20 copies/ml), measured at 6 months postpartum.
Proportion of infants HIV-positive at 2 and 6 months post-delivery. | At 2 months (62 days) and at 6 months (197 days) post-delivery.
  All exposed infants who tested positive by DNA-PCR at 6 - 8 weeks of age and at 6 months are included in analysis for "early" MTCT and "late" MTCT, respectively. Any infants testing positive at first/early DNA PCR are excluded for testing at 6 months of age.
Proportion of HIV-positive mothers retained in PMTCT care at 12 months post-delivery. | At 360 days (12 months) post-delivery
  Maternal retention is determined by evaluating for at least 1 clinic visit made for each 30-day period for the first 360 days postpartum. The proportion of women making at least 6 of 12 monthly appointments are designated retained; this proportion is calculated for each study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia A Sam-Agudu, MD, CTropMed, Principal Investigator — Institute of Human Virology, Nigeria; University of Maryland School of Medicine
Locations (1):
- Nadia Sam-Agudu, Abuja, Federal Capital Territory, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sam-Agudu NA, Cornelius LJ, Okundaye JN, Adeyemi OA, Isah HO, Wiwa OM, Adejuyigbe E, Galadanci H, Afe AJ, Jolaoso I, Bassey E, Charurat ME. The impact of mentor mother programs on PMTCT service uptake and retention-in-care at primary health care facilities in Nigeria: a prospective cohort study (MoMent Nigeria). J Acquir Immune Defic Syndr. 2014 Nov 1;67 Suppl 2:S132-8. doi: 10.1097/QAI.0000000000000331. PMID 25310119
- [Background] Cataldo F, Sam-Agudu NA, Phiri S, Shumba B, Cornelius LJ, Foster G. The Roles of Expert Mothers Engaged in Prevention of Mother-to-Child Transmission (PMTCT) Programs: A Commentary on the INSPIRE Studies in Malawi, Nigeria, and Zimbabwe. J Acquir Immune Defic Syndr. 2017 Jun 1;75 Suppl 2:S224-S232. doi: 10.1097/QAI.0000000000001375. PMID 28498193
- [Background] Sam-Agudu NA, Aliyu MH, Adeyemi OA, Oronsaye F, Oyeledun B, Ogidi AG, Ezeanolue EE. Generating evidence for health policy in challenging settings: lessons learned from four prevention of mother-to-child transmission of HIV implementation research studies in Nigeria. Health Res Policy Syst. 2018 Apr 17;16(1):32. doi: 10.1186/s12961-018-0309-x. PMID 29665809
- [Result] Al-Mujtaba M, Cornelius LJ, Galadanci H, Erekaha S, Okundaye JN, Adeyemi OA, Sam-Agudu NA. Evaluating Religious Influences on the Utilization of Maternal Health Services among Muslim and Christian Women in North-Central Nigeria. Biomed Res Int. 2016;2016:3645415. doi: 10.1155/2016/3645415. Epub 2016 Feb 24. PMID 27006944
- [Result] McCarthy E, Joseph J, Foster G, Mangwiro AZ, Mwapasa V, Oyeledun B, Phiri S, Sam-Agudu NA, Essajee S. Modeling the Impact of Retention Interventions on Mother-to-Child Transmission of HIV: Results From INSPIRE Studies in Malawi, Nigeria, and Zimbabwe. J Acquir Immune Defic Syndr. 2017 Jun 1;75 Suppl 2(2):S233-S239. doi: 10.1097/QAI.0000000000001364. PMID 28498194
- [Result] Sam-Agudu NA, Ramadhani HO, Isah C, Erekaha S, Fan-Osuala C, Anaba U, Adejuyigbe EA, Charurat M. The Impact of Structured Mentor Mother Programs on Presentation for Early Infant Diagnosis Testing in Rural North-Central Nigeria: A Prospective Paired Cohort Study. J Acquir Immune Defic Syndr. 2017 Jun 1;75 Suppl 2:S182-S189. doi: 10.1097/QAI.0000000000001345. PMID 28498188
- [Result] Sam-Agudu NA, Ramadhani HO, Isah C, Anaba U, Erekaha S, Fan-Osuala C, Galadanci H, Charurat M. The Impact of Structured Mentor Mother Programs on 6-Month Postpartum Retention and Viral Suppression among HIV-Positive Women in Rural Nigeria: A Prospective Paired Cohort Study. J Acquir Immune Defic Syndr. 2017 Jun 1;75 Suppl 2:S173-S181. doi: 10.1097/QAI.0000000000001346. PMID 28498187
- [Result] Odiachi A, Erekaha S, Cornelius LJ, Isah C, Ramadhani HO, Rapoport L, Sam-Agudu NA. HIV status disclosure to male partners among rural Nigerian women along the prevention of mother-to-child transmission of HIV cascade: a mixed methods study. Reprod Health. 2018 Mar 2;15(1):36. doi: 10.1186/s12978-018-0474-y. PMID 29499704
- [Result] Cornelius LJ, Erekaha SC, Okundaye JN, Sam-Agudu NA. A Socio-Ecological Examination of Treatment Access, Uptake and Adherence Issues Encountered By HIV-Positive Women in Rural North-Central Nigeria. J Evid Inf Soc Work. 2018 Jan-Feb;15(1):38-51. doi: 10.1080/23761407.2017.1397580. Epub 2017 Dec 13. PMID 29236624
- [Result] Sam-Agudu NA, Isah C, Fan-Osuala C, Erekaha S, Ramadhani HO, Anaba U, Adeyemi OA, Manji-Obadiah G, Lee D, Cornelius LJ, Charurat M. Correlates of facility delivery for rural HIV-positive pregnant women enrolled in the MoMent Nigeria prospective cohort study. BMC Pregnancy Childbirth. 2017 Jul 14;17(1):227. doi: 10.1186/s12884-017-1417-2. PMID 28705148
- [Result] Sam-Agudu NA, Odiachi A, Bathnna MJ, Ekwueme CN, Nwanne G, Iwu EN, Cornelius LJ. "They do not see us as one of them": a qualitative exploration of mentor mothers' working relationships with healthcare workers in rural North-Central Nigeria. Hum Resour Health. 2018 Sep 10;16(1):47. doi: 10.1186/s12960-018-0313-9. PMID 30200969
- [Derived] Odiachi A, Al-Mujtaba M, Torbunde N, Erekaha S, Afe AJ, Adejuyigbe E, Galadanci HS, Jasper TL, Cornelius LJ, Sam-Agudu NA. Acceptability of mentor mother peer support for women living with HIV in North-Central Nigeria: a qualitative study. BMC Pregnancy Childbirth. 2021 Aug 7;21(1):545. doi: 10.1186/s12884-021-04002-1. PMID 34364384
- [Derived] Odiachi A, Sam-Agudu NA, Erekaha S, Isah C, Ramadhani HO, Swomen HE, Charurat M, Cornelius LJ. A mixed-methods assessment of disclosure of HIV status among expert mothers living with HIV in rural Nigeria. PLoS One. 2020 Apr 30;15(4):e0232423. doi: 10.1371/journal.pone.0232423. eCollection 2020. PMID 32353036